CLINICAL TRIAL: NCT03888391
Title: 12 Month Open Extension Study of TNS for ADHD .
Brief Title: 12 Month Open Extension of TNS for ADHD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James McGough (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, James McGough, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMH R34 MH101282; R34MH101282 (NIH)
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Results first posted 2019-04-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; neuromodulation; trigeminal nerve stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open-label active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Active TNS (Experimental): Participants will receive trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for up to 12 months of this open-extension trial.
  Interventions: Device: Active TNS

INTERVENTIONS:
Device: Active TNS

SUMMARY:
Participants who exhibit sufficient ADHD symptom improvement in a prior study of active TNS will be invited to continue in a 12-month extension study, designed to collect additional data on long-term response and tolerability and to provide participants ongoing clinical benefit from treatment.

DETAILED DESCRIPTION:
Children, ages 8-12 years, participated in a 5 week double-blind, sham-controlled study of active Trigeminal Nerve Stimulation (TNS). Participants randomized to sham in the double-blind, were then invited into a 4-week open TNS trial. Participants who met positive response criteria to active TNS, either during the original double-blind study or the open-treatment followup, were invited to continue their TNS treatment in a 12-month open extension phase.

Participants who continued in the 12-month extension returned for study visits every 3 months to assess ongoing response and safety/tolerability data. Unless otherwise noted, baseline line assessments in the 12-month extension are taken from the final visit of the preceding active treatment trial, i.e. the visit at which positive response criteria were met.

ELIGIBILITY:
Inclusion Criteria:

* male and female children ages 8-13 with DSM-5 ADHD, and current presentation, as determined by KSADS and clinical interview
* received active TNS therapy in a previous trial and demonstrated a CGI-I score <= 2.
* parents able and willing to monitor proper use of the TNS device and complete all required rating scales
* parent and participants able to compete study rating scales and other measures in English

Exclusion Criteria:

* none

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-12-01; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. McGough, M.D., Principal Investigator — University of California, Los Angelesr; Sandra K. Loo, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active TNS
Started | 18
Completed | 3
Not Completed | 15
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Groups:
- Active TNS: Participants will receive trigeminal nerve stimulation (TNS) administered by the Monarch eTNS System nightly during sleep for up to 12 months of this open-extension trial.
  Active TNS:
Arm/Group | Active TNS
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.41 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
ADHD-Rating Scale Total Score [Mean (Standard Deviation); unit: score on a scale.] — A dimensional rating of ADHD symptoms, with scores ranging from 0 to 54, with higher scores signifying worse severity.
  score on a scale. | 16.56 (8.72)
Clinical Global Impression - Severity (CGI-S) [Count of Participants; unit: Participants] — A categorical measure of severity ranging from 1 ("Normal, not at all ill") to 7 ("Among the most seriously ill).
  Participants
    1 (Normal, not at all ill) | 0
    2 (Borderline ill) | 0
    3 (Mildly ill) | 2
    4 (Moderately ill) | 8
    5 (Markedly ill) | 8
    6 (Severely ill) | 0
    7 (Among the most extremely ill) | 0

OUTCOME MEASURES:

1. Primary Outcome: ADHD-IV Rating Scale (ADHD-RS)
Description: A dimensional rating of ADHD symptoms, with scores ranging from 0 to 54, with higher scores signifying worse severity.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Participants lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active TNS
Number analyzed (Participants) | 18
score on a scale
  Baseline | 19.06 (1.78)
  Month 3 | 16.56 (1.78)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 17.51 (2.45)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 15.55 (2.76)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 15.97 (3.72)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p = .20, Mixed Models Analysis; Time: F = 1.72, df = 1/34

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: Categorical measure indicating degree improved or not improved compared with global functioning at baseline in the preceding double-blind trial. The base CGI-I scale is a 7-point measure that requires the investigator to assess how much the condition has improved or worsened compared to baseline prior to initiation of treatment. Ratings are (1) very much improved; (2) much improved; (3) minimally improved; (4) no change; (5) minimally worse; (6) much worse; (7) very much worse. For purposes of analysis, the measure is dichotomized such that scores <= 2 signify "improved" and scores > 2 signify "not improved."
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants lost to follow up over time.
Measure: Count of Participants; unit: Participants
Arm/Group | Active TNS
Number analyzed (Participants) | 18
Participants
  Month 3: Improved | 16
  Month 3: Not Improved | 2
  Month 6: number analyzed (Participants) | 8
  Month 6: Improved | 8
  Month 6: Not Improved | 0
  Month 9: number analyzed (Participants) | 7
  Month 9: Improved | 7
  Month 9: Not Improved | 0
  Month 12: number analyzed (Participants) | 3
  Month 12: Improved | 3
  Month 12: Not Improved | 0

3. Secondary Outcome: Height
Description: A dimensional measure assessed in cm.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: cm.
Arm/Group | Active TNS
Number analyzed (Participants) | 18
cm.
  Baseline | 140.45 (2.12)
  Month 3 | 143.09 (2.11)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 144.20 (2.25)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 147.27 (2.32)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 148.37 (2.56)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p < .0001, Mixed Models Analysis; Time: F = 44.47, df = 1/33

4. Secondary Outcome: Weight
Description: A dimensional measure assessed in kg.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: kg.
Arm/Group | Active TNS
Number analyzed (Participants) | 18
kg.
  Baseline | 38.42 (3.20)
  Month 3 | 38.76 (3.20)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 39.37 (3.22)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 39.96 (3.23)
  Moth 12: number analyzed (Participants) | 3
  Moth 12 | 41.82 (3.28)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p = .0004, Mixed Models Analysis; Time: F = 15.74, df = 1/34

5. Secondary Outcome: Systolic Blood Pressure
Description: A dimensional measure assessed in mm Hg.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS
Number analyzed (Participants) | 18
mm Hg.
  Baseline | 109.06 (2.47)
  Month 3 | 108.72 (2.47)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 110.06 (3.50)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 109.79 (3.97)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 102.18 (5.42)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p = .60, Mixed Models Analysis; Time: F = .28, df = 1/34

6. Secondary Outcome: Diastolic Blood Pressure
Description: A dimensional measure assessed in mm Hg.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Active TNS
Number analyzed (Participants) | 18
mm Hg.
  Baseline | 61.89 (2.10)
  Month 3 | 64.33 (2.10)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 63.49 (3.01)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 64.40 (3.42)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 66.40 (4.70)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p = .32, Mixed Models Analysis; Time: F = 1.04, df = 1/34

7. Secondary Outcome: Pulse
Description: A dimensional measure assessed in heart beats per minute.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Population: Some participants were lost to follow up over time.
Measure: Least Squares Mean (Standard Error); unit: Heart beats per minute.
Arm/Group | Active TNS
Number analyzed (Participants) | 18
Heart beats per minute.
  Baseline | 81.56 (2.82)
  Month 3 | 80.78 (2.82)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 76.83 (3.64)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 79.76 (4.02)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 77.25 (5.23)
Statistical Analysis 1: Comparison: Active TNS; Outcomes fitted via a mixed model with time as a predictor; Test type: Superiority; p = .27, Mixed Models Analysis; Time: F = 1.27, df = 1/34

8. Other Pre Specified Outcome: Conners Global Index - Parent Report
Description: Parent completed dimensional rating of ADHD symptoms, with scores ranging from 0-30, and higher scores signifying more severe symptoms.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Conner Global Index - Teacher Report
Description: Teacher completed dimensional rating of ADHD symptoms, with scores ranging from 0-30, and higher scores indicating more severe symptoms.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Affective Reactivity Index (ARI-C) Child
Description: A child completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Affective Reactivity Index (ARI-P) Parent
Description: A parent completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Children's Sleep Habits Questionnaire (CSHQ)
Description: A parent completed 33-item scale to assess sleep related problems. Total scores range from 33 to 99, divided among 8 sub scales, with higher scores indicating more severe difficulties.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Multidimensional Anxiety Scale for Children (MASC) Child Report
Description: A child completed rating of child anxiety, with scores ranging from 0-300, and higher scores indicating greater severity.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Multidimensional Anxiety Scale for Children (MASC) Parent Report
Description: A parent completed measure of child anxiety, with scores ranging fro 0-300, and higher scores indicating greater severity.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Children's Depression Rating Scale - Revised (CDRS-R)
Description: A clinician completed dimensional measure of child mood symptoms, obtained from parent and child interview, with range of scores from 17 to 113, and higher scores indicating more severe depression. A score >= 40 suggests depression; scores <=28 define remission.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Behavior Rating Inventory of Executive Functioning (BRIEF)
Description: A parent completed rating of executive functioning. Comprises 5 sub scales that measure various measures of behavior and cognition. Raw scores for each measure are converted to T scores ranging from 28 to 103, with higher scores indicating greater difficulties.
Time Frame: Change over baseline, Month 3, Month 6, Month 9, Month 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, measured at 3, 6, 9, and 12 months.
Description: Adverse events were solicited via a structured side effects questionnaire and open inquiry, completed at each study visit.
Arm/Group | Active TNS
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 11/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TNS (N=18)
Trouble sleeping (Psychiatric disorders) | 3 (5)
Drowsy (General disorders) | 2 (2)
Hyperactive (Psychiatric disorders) | 6 (9)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomachache (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Frequent urination (Renal and urinary disorders) | 2 (3)
Increased appetite (General disorders) | 1 (1)
Difficulty finding words (Nervous system disorders) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Clenching teeth (Musculoskeletal and connective tissue disorders) | 1 (1)
Active suicidal ideation with plan and intent (Psychiatric disorders) | 0 (0) — Based on the Columbia - Suicide Severity Rating Scale (C-SSRS)
Active suicidal ideation with some intent (Psychiatric disorders) | 0 (0) — Based on the Columbia - Suicide Severity Rating Scale (C-SSRS)
Active suicidal ideation without intent (Psychiatric disorders) | 0 (0) — Based on the Columbia - Suicide Severity Rating Scale (C-SSRS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03888391/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT03888391/Prot_SAP_002.pdf